CLINICAL TRIAL: NCT02409173
Title: Effects of Noninvasive Positive Pressure Ventilation on Inflammatory Markers, Sleep, Pulmonary Function and HRQoL in Severe Obese Patients With Metabolic Syndrome Undergone to Bariatric Surgery. A Randomized Controlled Clinical Trial
Brief Title: NPPV on Inflammatory Markers and Sleep in Severe Obese Patients With Metabolic Syndrome Undergone to Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Centro Universitário de Anapolis (Other)
Responsible Party: Principal Investigator, Luis Vicente Franco de Oliveira, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 742.865/2014
Record Dates: First submitted 2015-03-24; First posted 2015-04-06 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Sleep disorders; Bariatric Surgery; Noninvasive ventilation; Inflammation; Quality of life
MeSH Terms: conditions — Metabolic Syndrome; Sleep Wake Disorders; Inflammation | interventions — Bariatric Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Noninvasive Ventilation and Surgery (Experimental): Noninvasive positive airway pressure flow generator device by full face or nasal mask and bariatric surgery.
  Interventions: Device: Noninvasive positive airway pressure flow generator device; Procedure: Bariatric Surgery
- Control Group (No Intervention)

INTERVENTIONS:
Device: Noninvasive positive airway pressure flow generator device — Noninvasive positive airway pressure flow generator device.
  Other Names: Noninvasive Positive Pressure Ventilation
  Arms: Noninvasive Ventilation and Surgery
Procedure: Bariatric Surgery — Standard Roux-en-Y gastric bypass
  Arms: Noninvasive Ventilation and Surgery

SUMMARY:
Obesity is currently one of the most serious public health problems. Its prevalence is increasing sharply in recent decades, even in developing countries, leading to global epidemiology condition. Metabolic syndrome (MS) consists of an association of metabolic and cardiovascular disorders including central obesity, insulin resistance, dyslipidemia and hypertension in the same patient. Obstructive sleep apnea (OSA) is a common clinical condition in more than 60% patients with MS. It is still controversial in the world scientific literature whether treatment of OSA with Noninvasive Positive Pressure Ventilation (NPPV) in severely obese patients with and without MS is effective. The NPPV effectively reverses hypoxemia in patients with OSA, therefore justified the hypothesis that NPPV will reduce insulin resistance, ghrelin and resistin and raise adiponectin levels in a group of severely obese individuals with and without MS undergoing bariatric surgery. Objectives: To investigate the effects of Noninvasive Positive Pressure Ventilation on inflammatory markers, sleep, pulmonary function, BMI reduction and health related quality of life in severe obese patients with and without metabolic syndrome undergone to bariatric surgery.

DETAILED DESCRIPTION:
Obesity is currently one of the most serious public health problems. Its prevalence is increasing sharply in recent decades, even in developing countries, leading to global epidemiology condition. Metabolic syndrome (MS) consists of an association of metabolic and cardiovascular disorders including central obesity, insulin resistance, dyslipidemia and hypertension in the same patient. Obstructive sleep apnea (OSA) is a common clinical condition in more than 60% patients with MS. It is still controversial in the world scientific literature whether treatment of OSA with Noninvasive Positive Pressure Ventilation (NPPV) in severely obese patients with and without MS is effective. The NPPV effectively reverses hypoxemia in patients with OSA, therefore justified the hypothesis that NPPV will reduce insulin resistance, ghrelin and resistin and raise adiponectin levels in a group of severely obese individuals with and without MS undergoing bariatric surgery. Objectives: To investigate the effects of Noninvasive Positive Pressure Ventilation on inflammatory markers, sleep, pulmonary function, BMI reduction and health related quality of life in severe obese patients with and without metabolic syndrome undergone to bariatric surgery. Methods/Design: Will participate severe obese patients with and without MS, screened from the Bariatric Surgery Service of Santa Casa de Sao Paulo. The inclusion criteria are patients with morbid obesity grade III, with an indication of bariatric surgery and who have agreed to the study, signing an informed consent. Subjects with BMI above 55 kg / m², clinically significant or mental health concerns unstable, an unrealistic target postsurgical weight and/or unrealistic expectations of the surgical treatment will be excluded. Patients will use the NPPV pre and post bariatric surgery. The evaluation protocol will consist of clinical history, vital signs, anthropometric data, clinical analysis of blood and adipose inflammatory markers, lung function tests, polysomnography, sleep scales, cardiovascular risk and quality of life questionnaires. Patients will be evaluated before and after bariatric surgery, 90, 180 and 360 days.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients aged 18 to 65 years,
* grade III severe obesity (BMI ≥ 40 kg/m2) or ≥ 35 kg/m2 with comorbidities,
* awaiting bariatric surgery,
* with documented history of conventional weight loss attempts having proven unsuccessful over time,
* sleep apnea history verified through polysomnography
* and if they are able to understand and agreement to participate in the study through a signed term of informed consent.

Exclusion Criteria:

* Any medical condition rendering surgery too risky,
* BMI above 55 kg/m2,
* unrealistic postoperative target weight and/or unrealistic expectations of surgical treatment,
* pregnancy,
* lactation or planned pregnancy within two years of potential surgical treatment,
* lack of safe access to abdominal cavity or gastrointestinal tract;
* abusive alcohol use or drug use,
* craniofacial abnormalities,
* undergoing active treatment of sleep apnea,
* cancer,
* any cardiorespiratory condition opposite indicate the surgical procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change in systemic immune response | Baseline immune response to 180 days.
  Systemic markers of inflammation through fasting blood samples biochemical indexes.
Change in systemic adipose inflammation response | Baseline adipose inflammation response to 180 days.
  Systemic markers of inflammation through biochemical indexes in visceral (omental, mesenteric) and subcutaneous adipose tissue depots.

SECONDARY OUTCOMES:
Prevalence of sleep disorders | 180 days
  Study sleep patterns through full standard polysomnography.
Changes in pulmonary function | 180 days
  Assess pulmonary function through pletysmography.
Changes in maximal ventilatory pressures | 180 days
  Assess maximal inspiratory and expiratory pressures through manovacuometry.
Changes in health related quality of life | 180 days
  Changes in quality of life through Short Form-36 and BAROS questionnaires.
Weight Loss | 180 days
  Body mass index reduction.

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Gastromed, Anápolis, Goiás
  - Department of Surgery of Santa Casa of Sao Paulo Medical School, São Paulo, São Paulo
  - Pulmonary Function Laboratory of Santa Casa of Sao Paulo Medical School, São Paulo, São Paulo